CLINICAL TRIAL: NCT04164394
Title: Efficacy of Probiotic I31 on Symptomatic Improvement in Patients With Lactose Intolerance
Brief Title: Effect of I31 Probiotic on Lactose Intolerance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Juarez de Mexico (Other Government)
Responsible Party: Principal Investigator, Nuria Pérez López, Digestive Physiology Lab Head, Hospital Juarez de Mexico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HJM 0431/18-R
Record Dates: First submitted 2019-11-11; First posted 2019-11-15 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-02

CONDITIONS: Lactose Intolerance
Keywords: Probiotic; Diarrhea; Abdominal pain; Flatulence
MeSH Terms: conditions — Lactose Intolerance; Diarrhea; Abdominal Pain; Flatulence

STUDY DESIGN:
Intervention Model Description: Allocation is 2:1 to probiotic and placebo arms
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo treatment (maltodextrin), once daily (u.i.d)
  Interventions: Other: Placebo
- Probiotic (Experimental): I31 probiotic formula (dietary supplement), consisting of 3 billion cfus of strains P. acidilactici CECT7483, L.plantarum CECT7484 and L.plantarum CECT7485, once daily (u.i.d)
  Interventions: Dietary Supplement: I31 Probiotic

INTERVENTIONS:
Other: Placebo — Placebo treatment (maltodextrin), once daily (u.i.d)
  Arms: Placebo
Dietary Supplement: I31 Probiotic — I31 probiotic formula (dietary supplement), consisting of 3 billion cfus of strains P. acidilactici CECT7483, L.plantarum CECT7484 and L.plantarum CECT7485, once daily (u.i.d)
  Arms: Probiotic

SUMMARY:
This randomized study evaluates the usefulness of the I31 probiotic formula, against placebo, in the treatment of symptoms of lactose intolerance.

DETAILED DESCRIPTION:
People with lactose intolerance are unable to fully digest the sugar (lactose) in milk. As a result, they may have diarrhea, abdominal pain, gas and bloating after eating or drinking dairy products. A deficiency of lactase - an enzyme produced in your small intestine - is usually responsible for lactose intolerance. Many people have low levels of lactase but are able to digest milk products without problems. In lactose intolerance, though, lactase deficiency leads to symptoms after eating dairy foods.

I31 is a probiotic formula composed of Pediococcus acidilactici strain CECT7483 and Lactobacillus plantarum strains CECT7484 and CECT7485, previously shown to improve intestinal sensitivity in patients with Irritable Bowel Syndrome (IBS). IBS is a functional intestinal disease in which recurrent abdominal pain is associated with defecation or a change in bowel habits, often accompanied by bloating. Given the overlap in symptoms between IBS and lactose intolerance, it is hypothesized that I31 formula could be beneficial for individuals with lactose intolerance.

ELIGIBILITY:
Inclusion Criteria:

* Subjects attending Hospital Juarez de Mexico with self-reported lactose intolerance, a minimum lactose intolerance symptom score of 6 points, 20ppm during the Lactose Hydrogen Breath Test (LHBT) and providing Informed Consent.

Exclusion Criteria:

* More than 10 ppm before ingestion of lactose in the Lactose Hydrogen Breath Test (LHBT). If such value was observed, the LHBT test was repeated on a 2nd day, and if >10ppm persisted, patient was excluded.
* BMI below 18 or above 40
* Subjects not accepting to maintain their dietary and physical activity pattern unchanged for the duration of the study
* Subjects with congenital lactase deficiency
* Pregnant or lactating women
* Significant gastrointestinal disease, such as inflammatory bowel disease, coeliac disease, chronic diarrhea or gastroparesis
* History of gastrointestinal surgery in the 6 months prior to inclusion
* History of intestinal perforation
* History of acute gastroenteritis, acute gastroenteritis or hospitalization in the 4 weeks prior to inclusion
* Substance abuse
* Untreated thyroid disorder
* Cancer
* Other severe diseases that in the doctor's opinion could interfere with the study
* Known allergy to any of the components in the treatments

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2019-05-13 (Actual); Primary Completion 2019-12-10 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Overall Symptoms Score | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  Total score of the "Symptoms Questionnaire for Lactose Malabsorption Screening" (Casellas et al. Dig Dis Sci 2009; 54:1059-65). Score ranges 0 to 50, where 50 represents maximum symptoms severity

SECONDARY OUTCOMES:
Abdominal Pain subscore | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  Abdominal pain Visual Analog Scale (VAS) subscore of the "Symptoms Questionnaire for Lactose Malabsorption Screening". Score ranges 0 to 10, where 10 represents maximum pain severity (Casellas et al. Dig Dis Sci 2009; 54:1059-65)
Vomiting subscore | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  Vomiting Visual Analog Scale (VAS) subscore of the "Symptoms Questionnaire for Lactose Malabsorption Screening". Score ranges 0 to 10, where 10 represents maximum vomiting severity (Casellas et al. Dig Dis Sci 2009; 54:1059-65)
Intestinal Sounds subscore | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  Intestinal Visual Analog Scale (VAS) sounds subscore of the "Symptoms Questionnaire for Lactose Malabsorption Screening". Score ranges 0 to 10, where 10 represents maximum intestinal sounds severity (Casellas et al. Dig Dis Sci 2009; 54:1059-65)
Flatulence subscore | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  Flatulence Visual Analog Scale (VAS) subscore of the "Symptoms Questionnaire for Lactose Malabsorption Screening". Score ranges 0 to 10, where 10 represents maximum flatulence severity (Casellas et al. Dig Dis Sci 2009; 54:1059-65)
Lactose Hydrogen Breath Test (LHBT) | 3 hours (performed after 25 gr lactose challenge, at baseline and after 8 weeks of intervention)
  LHBT test performed with 25 gr of lactose after an overnight fast. Measurements 10 minutes before lactose ingestion and 60, 120 and 180 minutes after lactose ingestion. CO2 (Carbon Dioxide) used as control. If more than 10ppm in the measurement before ingestion of lactose, and LHBT test was rescheduled and recommendations to avoid complex carbohydrates 24h before the test were repeated. Carbon dioxide (CO2) was measured and used to adjust breath sample for non-alveolar dilution of exhaled air.

CONTACTS AND LOCATIONS:
Overall Officials: Nuria Perez Lopez, MD, Study Director — Hospital Juarez de Mexico
Locations (1):
- Hospital Juarez de Mexico, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No